CLINICAL TRIAL: NCT02363751
Title: Prospective Phase II Study of Gemcitabine Plus Platinum Salt in Combination With Bevacizumab (Avastin®) for Metastatic Collecting Duct Carcinoma
Brief Title: Study of Gemcitabine+Platinum Salt+Bevacizumab Combination for Metastatic Collecting Duct Carcinoma (GETUG-AFU 24)
Acronym: BEVABEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1210; 2013-001179-19 (EudraCT Number)
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Collecting Duct Carcinoma (Kidney)
Keywords: Bellini; Metastatic; Chemotherapy; Bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Patients will be treated for a maximum of 6 (21 days) chemotherapy cycles (Gemcitabine+platinum salt+bevacizumab)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Patients will be treated for a maximum of 6 (21days) chemotherapy cycles (Gemcitabine+platinum salt+bevacizumab).
  In case of disease control (complete, partial or stable disease) treatment with bevacizumab 15 mg/Kg monotherapy every 21 days will be continued until disease progression or until the end of the 24 months of follow-up.
  Other Names: Avastin

SUMMARY:
Open-label, non-randomized, multicenter, phase II, single arm non comparative trial evaluating toxicity and efficacy of gemcitabine plus platinum salt in combination with bevacizumab in first-line setting in metastatic collecting duct carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be aged ≥18 years at the inclusion,
2. Patients with histologically confirmed metastatic collecting duct carcinoma (medullary accepted),
3. Available tumor samples for centralized reading by anatomopathologist,
4. Patients with or without nephrectomy,
5. At least one measurable lesion as per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1),
6. No prior chemotherapy nor anti-angiogenic drugs ; Prior adjuvant chemotherapy of localised disease admitted if it is stopped for more than 12 months at the inclusion date.,
7. No irradiation within 4 weeks before inclusion,
8. Absolute neutrophil counts (ANC) ≥1.5 x 10⁹/L,
9. Platelets ≥100 x 10⁹/L,
10. Hemoglobin ≥9 g/dL,
11. Hepatic function : AST and ALT ≤1.5 x ULN (≤4 x ULN in case of liver metastases); total bilirubin ≤1.5 x ULN; alkaline phosphatase <2 x ULN (≤4 x ULN in case of bone metastases),
12. Renal function : creatinine clearance ≥60 mL/min (MDRD calculation method) using cis-platin and >30 mL/min when using carboplatin,
13. Absence of proteinuria at baseline defined by <0.3 g of protein on urine sample or <0.5 g/24h on urine collection,
14. Prothrombin time (TP) or partial thromboplastin time (PTT) strictly less than 50% deviation from normal limits, of international normalized ratio (INR) strictly below 2, Note: The use of full-dose oral or parenteral anticoagulants as well as aspirin or clopidogrel is permitted as long as the INR or a PTT is within therapeutic limits (according to the medical standard of the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks at the time of study enrolment. Prophylactic use of anticoagulants is allowed.
15. ECG with normal or clinically insignificant as per investigator's judgement sinus rhythm,
16. ECOG Performance Status: 0 - 2,
17. Estimated life expectancy ≥12 weeks,
18. Patients who have received the information sheet, dated and signed the informed consent form,
19. Patient of child-bearing potential (for female patient: study entry after a menstrual period and a negative pregnancy test) must agree to use two medically acceptable methods of contraception (one for the patient and one for the partner) during the study and for 6 months after the last study treatment intake.
20. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures,
21. Patients affiliated to the Social Security System,

Exclusion Criteria:

1. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment,
2. Prior systemic treatment with chemotherapy or anti-angiogenic tyrosine kinase inhibitors such as axitinib, sunitinib, sorafenib, pazopanib, tivozanib, mTOR inhibitor (Temsirolimus or everolimus) and targeted VEGF drugs such as bevacizumab and VEGF trap,
3. Evidence of current spinal cord compression or leptomeningeal disease. Please note that patients with asymptomatic brain metastases are eligible,
4. Another histological type of renal cancer
5. Other malignancy within 3 years prior to inclusion (except basal cell carcinoma of the skin and/or in situ carcinoma of the cervix, and/or pT1/a bladder cancer),
6. Uncontrolled hypertension (≥160 mm Hg systolic and/or ≥90 mm Hg diastolic) while receiving medication,
7. Cardio-vascular disorders: congestive heart failure ≥ NYHA II, myocardial infarction or coronary artery bypass graft in the previous six months, ongoing severe or unstable angina,
8. LVEF value strictly less than 50%,
9. Current or recent (within 2 weeks of study enrolment) initiation of aspirin, clopidogrel), oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes,
10. History of clinically significant hemorrhagic or thromboembolic events in the past six months, or known inherited predisposition to bleeding or thrombosis or History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment; History of haemoptysis ≥ grade 2 (defined as ≥2.5 mL bright red blood per episode) within 1 month of study enrolment,
11. Patients who underwent, according to the investigator, a significant surgery such as but not limited to , abdominal, thoracic or neurologic surgery within 28 days before the first treatment administration or patient with a wound that is not already healed at the first treatment administration or patients who underwent a minor surgical procedure including placement of a vascular access device, within 2 days of the first study treatment,
12. Patients with active gastro-duodenal ulcer,
13. Patients with untreated bone fracture,
14. Peripheral neuropathy grade ≥2 (Toxicity Criteria-(CTCAE) v4.0),
15. Patients with active infection requiring intravenous antibiotics at the time of first study treatment,
16. In the opinion of the investigator, any evidence of other severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease), or any other acute or chronic medical condition that would make the patient inappropriate with this study,
17. Immunocompromised patients, including known seropositivity for human immunodeficiency virus (HIV),
18. Known hypersensitivity to any component of the investigational drugs or excipients,
19. Pregnant or lactating women,
20. Person deprived of their liberty or under judicial protection (including guardianship),
21. Patients with significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule or any condition which, in the opinion of the investigator, would preclude participation in this trial. Those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2020-03 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Composite endpoint : Objective response rate / Progression-free survival | 6 months
  The primary endpoint is composed of:
  * the objective response rate (CR or PR) according to RECIST criteria (V1.1) on the basis of measurable lesions defined at baseline,
  * the progression-free survival (PFS) rate at 6 months , PFS is defined as the absence of disease progression or death

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years max
  Progression-free survival (PFS) will be calculated from the date of the first dose of treatment to the date of progression or death (whichever comes first), or last date with no progression
The Overall Survival (OS) | 2 years max
  The Overall Survival (OS) will be calculated from the date of the first dose of treatment to the date of death (whatever the cause) or the date of last follow-up
The toxicity will be evaluated according to the NCI-CTC scale version 4.0 | 2 years max

CONTACTS AND LOCATIONS:
Overall Officials: Constance THIBAULT, Dr, Principal Investigator — Hôpital Européen Georges-Pompidou; Marc-Olivier TIMSIT, Dr, Study Chair — Hôpital Européen Georges-Pompidou
Locations (19):
- France (19):
  - Institut de Cancérologie de l'Ouest-Site Paul Papin, Angers
  - CHU Besançon, Besançon
  - Hôpital Saint André, Bordeaux
  - Centre François Baclesse, Caen
  - Hôpital Henri Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint-Louis, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Eugene Marquis, Rennes
  - Institut de cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - CHU Strasbourg - Hôpital Civil, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHR Bretonneau, Tours
  - Gustave Roussy, Cancer Campus, Grand Paris, Villejuif

REFERENCES:
- [Derived] Thibault C, Flechon A, Albiges L, Joly C, Barthelemy P, Gross-Goupil M, Chevreau C, Coquan E, Rolland F, Laguerre B, Gravis G, Pecuchet N, Elaidi RT, Timsit MO, Brihoum M, Auclin E, de Reynies A, Allory Y, Oudard S. Gemcitabine plus platinum-based chemotherapy in combination with bevacizumab for kidney metastatic collecting duct and medullary carcinomas: Results of a prospective phase II trial (BEVABEL-GETUG/AFU24). Eur J Cancer. 2023 Jun;186:83-90. doi: 10.1016/j.ejca.2023.03.018. Epub 2023 Mar 23. PMID 37054556